CLINICAL TRIAL: NCT06442514
Title: Enhancing an Intervention for Smokers With Chronic Pain Using IVR: A Randomized Clinical Trial of Smoking Cessation Counseling for Veterans
Brief Title: Pain and Smoking Study - Interactive Voice Response
Acronym: PASS-IVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 22-070
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Smoking; Pain; Smoking Cessation
MeSH Terms: conditions — Smoking; Pain; Smoking Cessation | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PASS-IVR (Experimental): An intervention that includes a proactive telehealth intervention combining evidence-based smoking cessation counseling augmented with behavioral approaches for coping with pain, and nightly Interactive Voice Response (IVR) calls. Veterans in PASS-IVR will also be offered 12-weeks of pharmacotherapy (e.g., NRT patches and one of two rescue methods such as nicotine lozenge or gum or varenicline) via telemedicine consult. The NRT dose and delivery route will be tailored to the number of cigarettes smoked per day (using an established protocol).
  Interventions: Behavioral: PASS-IVR
- Treatment as Usual (Other): Treatment as usual includes referral to the local smoking cessation clinic where Veterans may select a virtual individual or group based cognitive behavioral smoking cessation program with a trained psychology intern, postdoctoral fellow or staff psychologist. In conjunction, Veterans are encouraged but not required, by clinic staff, to connect with the VA Quitline and the VA's Annie text-messaging service to support their quit. Veterans are strongly encouraged to consider pharmacotherapy (e.g., NRT patches and one of two rescue methods such as nicotine lozenge or gum or varenicline). The NRT dose and delivery route will be tailored to the number of cigarettes smoked per day (using an established protocol - interested Veterans will be offered a telemedicine consult for this service
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: PASS-IVR — An intervention that includes a proactive telehealth intervention combining evidence-based smoking cessation counseling augmented with behavioral approaches for coping with pain, and nightly Interactive Voice Response (IVR) calls to report smoking status, pain, and pedometer-measured step counts, which the clinician will use to provide individualized feedback.
  Arms: PASS-IVR
Other: Treatment as Usual — Referral to the local smoking cessation VA clinic.
  Arms: Treatment as Usual

SUMMARY:
PASS2 aims to expand upon the recently completed study (PASS intervention), which tested the telephone delivery of a cognitive behavioral intervention (CBI). This study will use Interactive Voice Response (IVR) to optimize the intervention's effectiveness for smoking cessation among Veteran smokers with chronic pain.

DETAILED DESCRIPTION:
Veterans with chronic pain represent an important population in which to focus smoking cessation efforts. Smoking cessation among patients with chronic medical illnesses substantially decreases morbidity and mortality; yet, many patients (>50%) with chronic pain continue to smoke.

This study aims to:

1. Determine whether the existing integrated pain and smoking cessation (PASS intervention) augmented with IVR (PASS-IVR) is superior to treatment as usual (e.g., referral to standard VA smoking cessation clinic) enhanced with pharmacotherapy tele-consult (E-TAU) at 6 (primary endpoint) and 12 months on cigarette abstinence rates among non-depressed Veterans with chronic pain.
2. Determine whether PASS-IVR is superior to E-TAU at 6 (primary endpoint) and 12 months on pain interference.
3. Examine critical components of the intervention process to inform future program implementation.

ELIGIBILITY:
Inclusion Criteria:

* being an enrolled Veteran at VACHS;
* current tobacco use;
* willingness to make a quit attempt;
* significant chronic pain defined as >/=4 on the pain intensity portion of the Brief Pain Inventory (BPI) for more than 90 days.

Exclusion Criteria:

* active diagnosis of dementia or psychosis in medical record;
* severely impaired hearing or speech;
* lack of telephone access;
* enrollment in concurrent research study that might affect main outcomes of this study;
* terminal illness;
* non-English speaking;
* pregnancy;
* provider advising against exercise;
* planned surgeries; and
* clinically significant depressive symptoms (>10 PHQ-9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2026-03-30 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Cigarette Smoking Abstinence Rates | 6-month and 12-month follow-up
  In keeping with the SNRT recommendations for measuring abstinence, we will use prolonged abstinence as our main outcome and allow for a grace period around quit date. During the 6- and 12-month follow-ups, patients will be asked about prolonged abstinence, "Since [end of the grace period] have you ever smoked at least a part of a cigarette on each of 7 consecutive days?" and "After [end of the grace period] have you smoked any in each of 2 consecutive weeks".

SECONDARY OUTCOMES:
Point prevalent abstinence | 6-month and 12-month follow-up
  Patients will be asked whether they have smoked a cigarette, even a puff, in the past 7 days and, if no, will be asked whether they have smoked a cigarette, even a puff, in the past 30 days.
Pain intensity and pain-related functional interference | baseline, 6-months follow-up, and 12-months follow-up
  Pain intensity and interference will be assessed using the 11-item BPI. The BPI also assesses chronicity of pain and areas of the body with pain. The interference subscale has demonstrated adequate internal consistency and robust concurrent validity and responsivity among patients with chronic non-cancer pain. We have also added the PROMIS 8-item pain interference measure and the PROMIS 3-item pain intensity measure which has comparable responsiveness to BPI and excellent internal consistency (.96).

CONTACTS AND LOCATIONS:
Overall Officials: Lori Anne Bastian, MD MPH, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No